CLINICAL TRIAL: NCT02979925
Title: Improving Functions in Veterans With Post-Traumatic Peripheral Neuropathic Pain
Acronym: PTP-NP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2366-P; 1192133 (Other Grant/Funding Number: VA San Diego Healthcare System)
Record Dates: First submitted 2016-11-29; First posted 2016-12-02 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Neuropathic Pain
Keywords: neuropathic pain; TMS; nerve injury; transcutaneous magnetic stimulation
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active transcutaneous magnetic stimulation (Experimental): Active transcutaneous magnetic stimulation (TMS) at the target site of nerve damage/injury.
  Interventions: Device: Active Transcutaneous Magnetic Stimulation
- Sham transcutaneous magnetic stimulation (Sham Comparator): Sham TMS will consist of the same parameters as active, however, the subject will be shielded from the magnetic field of the coil.
  Interventions: Device: Sham Transcutaneous Magnetic Stimulation

INTERVENTIONS:
Device: Active Transcutaneous Magnetic Stimulation — Active transcutaneous magnetic stimulation (TMS) at the target site of nerve damage/injury.
  Other Names: TMS
  Arms: Active transcutaneous magnetic stimulation
Device: Sham Transcutaneous Magnetic Stimulation — Sham TMS will consist of the same parameters as active, however, the subject will be shielded from the magnetic field of the coil.
  Other Names: TMS
  Arms: Sham transcutaneous magnetic stimulation

SUMMARY:
The proposed study will set the foundation for future multi-center studies. To validate tMS as a non-contact and non-invasive pain treatment option for reducing pain in Veterans with PTP-NP and improving their overall functions.

DETAILED DESCRIPTION:
This study will only be conducted at the VA hospital in San Diego.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Subject is willing and able to comply with scheduled visits, treatment plan, daily pain, sleep and all study related assessments and procedures
* Subjects must be literate in the language used in the assessments and pain diary
* Veterans (men or women) of any race or ethnicity who are at least 18 years of age
* Female subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 7 days after the last session of the assigned treatment

  * A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active
* Subject must have chronic peripheral neuropathic pain present for more than 4 months after a traumatic or surgical event per medical history, this may include, for example:

  * motor vehicle accident
  * fall
  * sports injury
  * knee or hip replacement
  * hernia repair
  * thoracotomy
  * mastectomy
  * focal/localized burns or crush injury
* In addition, to be eligible for inclusion in the study, all subjects must:

  * have an average daily Numerical Pain Rating Scale (NPRS) score >3 during B1; and
  * have a spontaneous pain intensity >30 on 0-100 Mechanical Visual Analogue Scale (M-VAS) to be eligible for randomization
* Must have their implicated peripheral nerve(s) identified
* Must meet criteria for neuropathic pain assessment to meet eligibility for the study [46]. Pain distribution across a nerve territory and history indicates relevant lesion or disease plus criteria listed in a and/or b
* (A): At least one negative or positive sensory sign or symptom confined to innervation territory of the lesioned nervous structure. Examples of negative or positive signs or symptoms include:

  * Burning, stabbing or tingling sensation/pain
  * Numbness/paresthesia
  * Cold, heat or pressure
  * Hyperalgesia or allodynia
  * Hypoesthesia
  * Increased or decreased sharp sensation (e.g., pinprick testing)
  * Decreased vibration/vibratory sensation
* (B): Prior diagnostic tests confirming lesion or disease explaining neuropathic pain (Nerve conduction studies, EMG, skin or nerve biopsy). Documentation of affected nerve(s) indicating that the subject's pain is of neuropathic origin and is a result of injury/trauma to the affected/implicated nerve(s).

Exclusion Criteria:

Subjects presenting with ANY of the following will NOT be included in the study:

* Subjects with neuropathic pain due to:

  * diabetic peripheral neuropathy
  * post herpetic neuralgia
  * Human Immunodeficiency Virus
  * chemo/anti-viral therapy
  * trigeminal neuralgia
  * carpal tunnel syndrome
  * subjects whose post-traumatic neuropathic pain is categorized as central (e.g., spinal cord injury) rather than peripheral
* Subjects with pain due to Complex Regional Pain Syndrome (CRPS, Type I or Type II)
* Phantom limb pain after amputation. However, subjects with stump pain and phantom sensation but no phantom pain will not be excluded
* Subjects with skin conditions in the affected dermatome that in the judgment of the investigator can interfere with evaluation of the neuropathic pain condition
* Subjects with other pain such as lumbar or cervical radiculopathy that may confound assessment or self-evaluation of the peripheral neuropathic pain

  * subjects with significant somatic pain at the site of their trauma that may confound assessment or self-evaluation of their neuropathic pain
* Any subject considered at risk of suicide or self-harm based on investigator judgment and/or the details of a risk assessment
* Use of prohibited medications in the absence of appropriate washout periods
* Participation in any other clinical trial within the 30 days prior to screening and/or during participation in this study
* Subjects with a history of a cardiac arrhythmia that has led to the placement of a cardiac pacer or defibrillator will be excluded from the study
* Pregnant females and females of childbearing potential not using highly effective contraception or not agreeing to continue highly effective contraception during the study
* Subjects with a current diagnosis of DSM-IV-TR Axis I disorder, including, for example:

  * schizophrenia
  * bipolar disorder
  * other psychotic disorders such as schizoaffective disorder and delusion disorder
  * somatoform disorders or factitious disorders
  * bipolar disorders, even if controlled or stable
  * alcohol or substance related disorders in the past 2 years
  * however, diagnoses of Generalized Anxiety Disorder (GAD) or major depression (MDD) that is clinically stable are allowed
* Subjects with pending Worker's Compensation, Worker's Compensation, civil litigation or disability claims pertinent to the subject based upon trauma

  * current involvement in out-of-court settlements for claims pertinent to subject's trauma
  * subjects with fully resolved litigation and compensation claims can participate
* Subjects who have previously received either transcranial or transcutaneous magnetic stimulation therapy in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yick Leung, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from October 2016 to June 2018 at the VA San Diego Medical Center.
Period: Overall Study
Arm/Group | Active Transcutaneous Magnetic Stimulation | Sham Transcutaneous Magnetic Stimulation
Started | 28 | 29
Completed | 28 | 23
Not Completed | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Transcutaneous Magnetic Stimulation | Sham Transcutaneous Magnetic Stimulation | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.11 (17.02) | 50.78 (14.04) | 52.61 (15.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 25 | 20 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 24 | 16 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 19 | 14 | 33
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 23 | 51
Spontaneous Pain Score [Mean (Standard Deviation); unit: score on a scale] — Spontaneous pain level was measured using a sliding algometer, known as the Mechanical Visual Analog Scale (M-VAS). The device has been well validated, and is anchored at the left by "no pain sensation" and at the right by "the most intense pain sensation imaginable." The corresponding length of the red bar with a scale from 0 to 100, which can be read on the back by the tester, represents the subject's intensity of pain. 0 represents "no pain sensation" and 100 represents "the most intense pain sensation imaginable." A lower value indicates a better outcome with lower levels of pain reported.
  score on a scale | 53.52 (21.01) | 49.13 (22.61) | 50.44 (22.69)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Spontaneous Pain Scores
Description: Spontaneous pain rating: Spontaneous pain level will be measured by using a sliding algometer, known as the Mechanical Visual Analog Scale (M-VAS). The device has been well validated, and is anchored at the left by "no pain sensation" and at the right by "the most intense pain sensation imaginable." The corresponding length of the red bar with a scale from 0 to 100, which can be read on the back by the tester, represents the subject's intensity of pain. 0 represents "no pain sensation" and 100 represents "the most intense pain sensation imaginable." A lower value indicates a better outcome with lower levels of pain reported.
Time Frame: Assessed during each of the subject's baseline visit, 1 week post treatment visit, and 4 weeks post treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcutaneous Magnetic Stimulation | Sham Transcutaneous Magnetic Stimulation
Number analyzed (Participants) | 28 | 23
score on a scale
  Baseline | 53.52 (21.01) | 49.13 (22.61)
  1 week post treatment | 41.41 (30.09) | 46.17 (26.54)
  4 weeks post treatment | 38.92 (29.16) | 37.52 (30.01)
Statistical Analysis 1: Comparison: Active Transcutaneous Magnetic Stimulation vs Sham Transcutaneous Magnetic Stimulation; Test type: Superiority; p = 0.246, Mixed Models Analysis

2. Secondary Outcome: Evaluation of Evoked Pain Scores: Stroking
Description: Stroking evoked pain will be assessed by gently moving a paintbrush over the site of PTNP. The patients will be asked if pain is felt. If so, the intensity of pain will be rated on a scale known as the Mechanical Visual Analog Scale (M-VAS). The device has been well validated, and is anchored at the left by "no pain sensation" and at the right by "the most intense pain sensation imaginable." The corresponding length of the red bar with a scale from 0 to 100, which can be read on the back by the tester, represents the subject's intensity of pain. 0 represents "no pain sensation" and 100 represents "the most intense pain sensation imaginable." A lower value indicates a better outcome with lower levels of pain reported.
Time Frame: Assessed during each of the subject's baseline visit, 1 week post treatment visit, and 4 weeks post treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcutaneous Magnetic Stimulation | Sham Transcutaneous Magnetic Stimulation
Number analyzed (Participants) | 28 | 23
score on a scale
  Baseline | 33.55 (31.07) | 24.78 (25.59)
  1 week post treatment | 30.74 (23.78) | 20.04 (24.10)
  4 weeks post treatment | 26.92 (21.90) | 21.35 (25.21)
Statistical Analysis 1: Comparison: Active Transcutaneous Magnetic Stimulation vs Sham Transcutaneous Magnetic Stimulation; Test type: Superiority; p = 0.651, Mixed Models Analysis

3. Secondary Outcome: Evaluation of Evoked Pain Scores: Von Frey
Description: Punctate evoked pain will be conducted by gently pressing a 5.18 von Frey monofilament against the site of PTNP. The patients will be asked if pain is felt. If so, the intensity of pain will be rated on a scale known as the Mechanical Visual Analog Scale (M-VAS). The device has been well validated, and is anchored at the left by "no pain sensation" and at the right by "the most intense pain sensation imaginable." The corresponding length of the red bar with a scale from 0 to 100, which can be read on the back by the tester, represents the subject's intensity of pain. 0 represents "no pain sensation" and 100 represents "the most intense pain sensation imaginable." A lower value indicates a better outcome with lower levels of pain reported.
Time Frame: Assessed during each of the subject's baseline visit, 1 week post treatment visit, and 4 weeks post treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcutaneous Magnetic Stimulation | Sham Transcutaneous Magnetic Stimulation
Number analyzed (Participants) | 28 | 23
score on a scale
  Baseline | 53.97 (27.04) | 43.13 (26.84)
  1 week post treatment | 46.89 (25.98) | 36.22 (26.22)
  4 weeks post treatment | 49.27 (24.72) | 38.26 (23.08)
Statistical Analysis 1: Comparison: Active Transcutaneous Magnetic Stimulation vs Sham Transcutaneous Magnetic Stimulation; Test type: Superiority; p = 0.902, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from first treatment to 4 weeks after the last treatment.
Arm/Group | Active Transcutaneous Magnetic Stimulation | Sham Transcutaneous Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/23

LIMITATIONS AND CAVEATS:
One limitation of this study is small sample size. In addition, the location of nerve damage (whether it is extremities or truncal region) could be a confounding factor for the effectiveness of the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT02979925/Prot_SAP_000.pdf